CLINICAL TRIAL: NCT03250013
Title: Long-term Effects of Medication for Attention Deficit Hyperactivity Disorder (ADHD) in Children and Adolescents on Cognition, Everyday Function and Quality of Life
Brief Title: Long-term Effects of Medication for ADHD
Acronym: LMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMA trial Goteborg
Record Dates: First submitted 2017-08-04; First posted 2017-08-15 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Children and adolescents with ADHD (Experimental): Children and adolescents medicating for ADHD of any subtype (presentation) with comorbidities
  Interventions: Drug: ADHD medications

INTERVENTIONS:
Drug: ADHD medications

SUMMARY:
Single-centre open-label prospective study, enrolling 127 children and adolescents aged 6-17 years, who receive medication for ADHD of any subtype (presentation). Long-term results are evaluated with tests of ADHD symptoms (Qb-test), intellectual ability (Wechsler scales; WISC), adaptive functioning (Vineland scale), everyday functioning (Weiss Functional Impairment Scale; WFIRS), and quality of life (Child Health and Illness Profile-Child Edition Scale; CHIP-CE) during 24 months of ADHD treatment.

DETAILED DESCRIPTION:
Single-centre open-label prospective study, including 127 subjects over a period of 2 years. Children and adolescents (6-17 years) who have been diagnosed with ADHD will be enrolled and followed during 24 months of ADHD treatment.

Screening assessments include medical, neurodevelopmental and psychiatric history, clinical evaluation and definition of the ADHD diagnosis and its subtypes or presentations (according to Diagnostic and Statistical Manual (DSM) IV and DSM 5), ADHD symptom severity and global functional impairment (by the investigator-rated ADHD Rating Scale-IV (ADHD-RS-IV) and Clinical Global Impression Scale-Severity and Improvement; CGI-S and CGI-I), comorbidities (by the Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) clinical interview), intellectual ability (by the WISC test), and general level of functioning (by the Vineland interview). Subjects previously assessed and diagnosed will be re-assessed at the screening visit to ascertain a current evaluation and definition of these parameters.

At baseline, a Qb-test and an assessment of symptom severity and global functional impairment will be made by the investigator-rated ADHD-RS-IV and CGI-S, everyday functioning by parent-rated WIFRS, and quality of life by parent-rated CHIP-CE. An adverse events report will be collected by interview with open-ended questions. Assignment to treatment will be individualized according to clinical picture and patient preference.

At subsequent visits (1, 2, 3, 6, 12, 18 and 24 months) the following assessments will be performed: Investigator-rated ADHD-RS-IV, CGI-S, Clinical Global Impression-Improvement (CGI-I) scales for symptom severity, global functional impairment and improvement. Adverse event report. Compliance assessment through pill count. Assessment of comorbidity status according to DSM-IV and DSM 5 checklist/interview.

A Qb-test will be performed at the 1 and 12 month visits. Everyday functioning and quality of life will be assessed by parent-rated WIFRS and CHIP-CE scales at the 12 and 24 month visits.

Duration of study treatment per subject is 24 months. Medication dosage is 1-3 doses daily as needed to optimize symptom control. Medications (methylphenidate, amphetamine, atomoxetine) will be provided by the pharmacy according to routines in standard clinical treatment.

For cluster analysis of Qb-test results, retrospective data from at least 50 patients previously diagnosed at our clinic will be added to the data from the subjects participating in the prospective study, to increase sample size to ascertain sufficient power for subgroup (cluster) analysis.

Safety evaluations Adverse event (AE) reports will be collected at all visits through open-ended questions. Vital signs (height, weight, blood pressure, pulse) will be assessed at all visits. AE severity should be graded: Mild, Moderate or Severe, and all AEs must be followed until an outcome is known, ensuring the subject's safety. All AEs will be recorded in the subject's medical records and in the Clinical Report Form (CRF), and also reported to the Medical Products Agency according to local regulations.

Study population Approximately 100 subjects from our centre will be enrolled in the prospective study.

Retrospective data for the cluster analysis will be collected from at least 50 patients previously diagnosed at our centre.

ELIGIBILITY:
Inclusion Criteria:

1. Children 6-17 years of age
2. Clinical diagnosis ADHD of any subtype and DSM 5 presentation
3. Intellectual ability in the normal range, according to Wechsler tests and clinical judgment
4. Subjects treated with ADHD medication will have a wash-out period prior to Qb-test at baseline, of 1 week for methylphenidate or amphetamine, 2 weeks for atomoxetine

Exclusion Criteria:

1. Physical or psychological limitation making Qb-test unsuitable.
2. Cardiovascular disease, seizures or other unstable medical conditions that might increase the risk for the subject.
3. Bipolar Disorder, Conduct Disorder, Psychosis, severe autism or other severe comorbid or medical conditions that in the investigator's opinion would make study participation unsuitable.
4. Concomitant medications (allowed at investigator's discretion), must be recorded in the subject's medical records and the CRF.
5. Substance use.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change in CGI - (S and I) | 0, 1, 2, 3, 6, 12, 18 and 24 months
  Investigator-rated clinical global impression scale - severity and improvement

SECONDARY OUTCOMES:
ADHD Rating Scale | 0, 1, 2, 3, 6, 12, 18 and 24 months
  Clinician-rated ADHD symptom scale
Qb-test | 0, 1 and 12 months
  Computerized ADHD-test
WISC-IV | 0 and 12 months
  Wechsler Intelligence Scale for Children
Vineland scale | 0 and 12 months
  Vineland parent interview of functioning
Weiss Functional Impairment Scale (WFIRS) | 0, 12 and 24 months
  Parent-rated function scale
Child Health and Illness Profile - Child Edition (CHIP-CE) | 0, 12 and 24 months
  Parent-rated quality of life scale

CONTACTS AND LOCATIONS:
Overall Officials: Mats Johnson, MD, PhD, Principal Investigator — Child Neuropsychiatry Unit, Sahlgrenska University Hospital, Gothenburg, Sweden
Locations (1):
- Child Neuropsychiatry Unit, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No